CLINICAL TRIAL: NCT04261062
Title: Validity Test of Wearable Continuous Blood Pressure Measuring System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2019-0080
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Patients in Surgical Intensive Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject: Patients in surgical intensive unit

SUMMARY:
1. Purpose of Research For the feasibility test of a wearable blood pressure measuring device, biometric data of patients in surgical intensive care is simultaneously obtained and stored from the device and a patient monitor.
2. Overview of Research Design This research is simply to obtain and store the data: 1) invasive arterial blood pressure measured with a patient monitor from one wrist, and 2) multi-wavelength photoplethysmography and pressure signal measured with the developed wearable device from the other wrist.
3. Medical Device for Clinical Trial Patient monitor (IntelliVue MX700, Philips, NED) and wearable blood pressure measuring device
4. Target Recruiting Number of Participants Considering the expected patient number in intensive care and 10% dropout rate during the research period, the target recurring number of participants is 220.
5. Criteria of Participant Inclusion

   1. Adult patient in surgical intensive care of Severance Hospital
   2. Voluntarily agreed to participate the research and not included to the exclusion criteria
6. Criteria of Participant Exclusion

   1. Patient with occlusive peripheral arterial disease
   2. Patient with cardiovascular disease of serious arrhythmia except atrial fibrillation
   3. Patient administered high-dose of pressor agent over 15 mcg/min
   4. Patient who is not available for measurement of invasive arterial blood pressure
   5. Patient who is not available to wear an wearable device on the wrist
   6. Pregnant woman, minor
7. Evaluation Parameter

   1. Systolic and diastolic blood pressure, which extracted in mmHg unit from the continuous blood pressure output of patient monitor.
   2. Blood pressure, which estimated by the signal analysis of multi-wavelength photoplethysmography and pressure signal measured with the wearable device.
8. Data Analysis and Statistical Methods

   1. From the multi-wavelength photoplethysmography and multi-channel pressure signal measured, continuous blood pressure will be estimated through the hemodynamic model and machine learning model.
   2. For the machine learning model, the data obtained will be divided into the training data and evaluation data, with the ratio of 80% and 20%.
   3. In order to evaluate the accuracy of the estimated blood pressure, the invasive arterial blood pressure will be considered as the reference blood pressure. Between the estimated blood pressure and the reference blood pressure, the correlation and root mean square error (RMSE) will be calculated.

DETAILED DESCRIPTION:
1. Recruit participants.
2. Explain the research purpose and details, and then have the participant sign the consent form.
3. Before starting the measurement, gather the participant's information such as age, length, and weight.
4. Measure noninvasive blood pressure in both arms. Compared to the blood pressure in the arm where inserted a catheter, confirm if difference of systolic or diastolic blood pressure in the other side of arm is not more than 10%.
5. Wear the wearable device on the opposite wrist from the catheter-inserted.
6. For 10 minutes, simultaneously obtain the data: 1) invasive arterial blood pressure measured with a patient monitor, and 2) multi-wavelength photoplethysmography and pressure signal measured with the developed wearable device.
7. For accuracy of data acquisition, repeat twice the procedure 5-7 by performing it in the morning and in the afternoon with the 5 hours interval.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient in surgical intensive care of Severance Hospital
2. Voluntarily agreed to participate the research and not included to the exclusion criteria

Exclusion Criteria:

1. Patient with occlusive peripheral arterial disease
2. Patient with cardiovascular disease of serious arrhythmia except atrial fibrillation
3. Patient administered high-dose of pressor agent over 15 mcg/min
4. Patient who is not available for measurement of invasive arterial blood pressure
5. Patient who is not available to wear an wearable device on the wrist
6. Pregnant woman, minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in surgical intensive care
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Title quality of pulsewave | 2 years

SECONDARY OUTCOMES:
User Comfortability | 2 years
  Abnormal symptoms or discomforts reported in wearing device

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of Anesthesiology and Pain Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes DJ, Babbs CF, Geddes LA, Bourland JD. Measurements of Young's modulus of elasticity of the canine aorta with ultrasound. Ultrason Imaging. 1979 Oct;1(4):356-67. doi: 10.1177/016173467900100406. No abstract available. PMID 575833
- [Background] Liu J, Yan BP, Dai WX, Ding XR, Zhang YT, Zhao N. Multi-wavelength photoplethysmography method for skin arterial pulse extraction. Biomed Opt Express. 2016 Sep 27;7(10):4313-4326. doi: 10.1364/BOE.7.004313. eCollection 2016 Oct 1. PMID 27867733
- [Background] Guanqun Zhang, Cottrell AC, Henry IC, McCombie DB. Assessment of pre-ejection period in ambulatory subjects using seismocardiogram in a wearable blood pressure monitor. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:3386-3389. doi: 10.1109/EMBC.2016.7591454. PMID 28269030
- [Background] Corino VD, Lombardi F, Mainardi LT. Blood pressure variability in patients with atrial fibrillation. Auton Neurosci. 2014 Oct;185:129-33. doi: 10.1016/j.autneu.2014.08.002. Epub 2014 Aug 17. PMID 25183309
- [Background] Michard F. Changes in arterial pressure during mechanical ventilation. Anesthesiology. 2005 Aug;103(2):419-28; quiz 449-5. doi: 10.1097/00000542-200508000-00026. PMID 16052125
- [Background] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265